CLINICAL TRIAL: NCT04688684
Title: The Emirates Heart Health Project: A Stepped-wedge Cluster Randomized-controlled Trial of a Family-based Health Coach Guided Dietary and Exercise Intervention for Reducing Weight and Cardiovascular Risk in Overweight and Obese Adult Nationals of the United Arab Emirates.
Brief Title: The Emirates Heart Health Project: A Family-based Diet and Exercise Intervention in Obese and Overweight Patients
Acronym: EHHP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Jeffrey King, Assistant Professor, United Arab Emirates University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: G00003405
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Overweight and Obesity; Cardiovascular Risk Factor
Keywords: overweight; obesity; cardiovascular risk; hypertension; hyperlipidemia; hemoglobin A1c
MeSH Terms: conditions — Overweight; Obesity; Hypertension; Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family-based intervention (Experimental): These participants will undergo the health coach based intervention with fitness tracker and diet changes, which will be delivered to all family members who meet the inclusion criteria and are enrolled in the study.
  Interventions: Behavioral: Family-based diet and exercise intervention

INTERVENTIONS:
Behavioral: Family-based diet and exercise intervention — The participants will meet together weekly as a family unit to receive education and planning to implement diet and lifestyle changes under the supervision of a health coach. This coach will also be available during the week by telephone or messaging for additional individualized support if needed.

SUMMARY:
Data from Abu Dhabi's Department of Health document that the leading cause of death among the population of the emirate of Abu Dhabi is cardiovascular disease (CVD). Even with significant investment of time and resources, this has not improved over time. CVD was the cause of death in over 39% of deaths occurring in patients above 45 years of age. In those older than 60 years of age, CVD causes more deaths than cancer, respiratory diseases, and infectious disease combined.

Eating an unhealthy diet is the leading risk factor for CVD-related deaths and one study estimated that the current diet accounted for 72% of CVD-related deaths in the United Arab Emirates (UAE). Interestingly, the limited intake of whole grains was associated with 22% of CVD-related deaths in the UAE. Other risk factors include consumption of processed meat, red meat, and sugar sweetened beverages.

Despite recognition of what constitutes healthy diet and exercise practices by survey participants, barriers exist to lifestyle change. In one UAE study of patients with type 2 diabetes, only 3% of the 390 individuals surveyed met numerous guidelines' weekly recommendations for 150 minutes of moderate intensity aerobic activity or 90 minutes of vigorous aerobic activity. The most common reasons given in that study for not exercising included cultural reasons (29.2%), "exercise is boring" (20.3%), and lack of family support (4.1%). Widespread availability and access to outpatient dieticians has not lowered rates of obesity, overweight, and cardiovascular disease risk factors.

To the investigators' knowledge, this would be the first study investigating the effect of a package of family based lifestyle interventions guided by a health coach. This package of interventions would be supported by technology such as a smartphone application to record dietary intake and the use of wearable fitness trackers to track physical activity. The nationals of the UAE (called Emiratis),have retained traditional cultural values, including strong ties to extended family, which may lead to better adherence to family based rather than individual appointments and interventions, which could lower CVD risk.

DETAILED DESCRIPTION:
Introduction In the past century, non-communicable diseases (NCDs) replaced infectious diseases as the leading cause of death worldwide. Despite concerted efforts by nations and health systems, NCDs continue to contribute to the deaths of millions each year. A growing body of literature suggests that these diseases may be associated with modern lifestyles which include reduced physical activity and an increased intake of calorie-dense nonnutritive foods leading to obesity (1,2) and overweight (3). Elevated body-mass-index (BMI) is associated with increased risk of cardiovascular disease (4, 5) as well as cancer (6). These trends have been documented in the United Arab Emirates (UAE), as well as in the specific region of this study, the emirate of Abu Dhabi (7, 8).

Existing knowledge Data from Abu Dhabi's Department of Health document that the leading cause of death among the population of the emirate of Abu Dhabi is cardiovascular disease (CVD) (7, 8). Even with significant investment of time and resources, this has not improved over time. CVD was the cause of death in over 39% of deaths occurring in patients above 45 years of age. In those older than 60 years of age, CVD causes more deaths than cancer, respiratory diseases, and infectious disease combined. (7) Eating an unhealthy diet is the leading risk factor for CVD-related deaths and one study estimated that the current diet accounted for 72% of CVD-related deaths in the United Arab Emirates (UAE). Interestingly, the limited intake of whole grains was associated with 22% of CVD-related deaths in the UAE. Other risk factors include consumption of processed meat, red meat, and sugar sweetened beverages (5).

Despite recognition among the population of the UAE regarding what constitutes healthy diet and exercise practices, barriers exist to lifestyle change. In one study of patients in the UAE with type 2 diabetes, only 3% of the 390 individuals surveyed met numerous guidelines' weekly recommendations for 150 minutes of moderate intensity aerobic activity or 90 minutes of vigorous aerobic activity. The most common reasons given in that study for not exercising included cultural reasons (29.2%), "exercise is boring" (20.3%), and lack of family support (4.1%).

Widespread availability and access to outpatient dieticians has not lowered rates of obesity, overweight, and cardiovascular disease risk factors.

Despite access to appointments on an individual basis, rates of obesity, overweight, and CVD risk factors have not improved.

To the investigators' knowledge, this would be the first study in the UAE investigating the effect of a package of family based lifestyle interventions guided by a health coach. This package of interventions would be supported by technology such as a smartphone application to record dietary intake and the use of wearable fitness trackers to track physical activity. The nationals of the UAE (called Emiratis),have retained traditional cultural values, including strong ties to extended family, which may lead to better adherence to family based rather than individual appointments and interventions, which could lower CVD risk.

Comparators The current practice in Kanad Hospital is to refer individual overweight and obese Emiratis to dieticians for co-management. In a stepped-wedge study, pre-intervention assessments of weight and cardiovascular risk of participants serve as a control, and will reflect the effects of current practice while clusters are awaiting the health coach led intervention. Once each family cluster has completed the intervention, the same assessments will be repeated and compared using a mixed effects model. The effectiveness of the Emirates Heart Health Program (EHHP) intervention will be measured. If found to have significant benefit, this package of interventions may be used in wider practice and influence both health insurance coverage and allocation of government resources.

Objectives Research hypothesis: The Emirates Heart Health Program (EHHP) is a family-based intervention using a health coach assisted by technological aids to make changes to participants' diet and exercise. This intervention package significantly reduces cardiovascular risk factors in the care of obese and overweight patients in the emirate of Abu Dhabi, United Arab Emirates.

Study Objectives:

Primary objective: to determine if the EHHP reduces of weight and BMI in obese and overweight Emiratis.

Secondary objectives: to determine in obese and overweight Emiratis, if the EHHP leads to:

* Reduction in systolic blood pressure Reduction in diastolic blood pressure
* Reduction in hemoglobin A1c
* Reduction in LDL cholesterol, total cholesterol, and triglycerides
* Increase in HDL.

Study setting: Study recruitment will take place in the outpatient clinics of Kanad Hospital in the emirate of Abu Dhabi, United Arab Emirates. 51.3% of patients visiting the hospital clinics in 2021 were Emirati.

Methods and analysis Trial design The EHHP is a family-cluster randomized stepped-wedge clinical trial, where the cluster units of randomization will be extended families. The order of family-clusters entering the intervention will be selected through randomization.

Interventions A health coach will deliver the program in the family's home, with 16 teaching and discussion sessions. These weekly sessions have used the DPP framework, and have been translated from English to Arabic and adapted to suit the Emirati culture and customs. The material for each session is largely scripted for standardization. Between sessions, the health coach will review the weight, dietary logbook, and wearable fitness tracker exercise records of each participant and provide additional support if needed. Assessment of height, weight, blood pressure and serum studies will be obtained in the outpatient clinic at scheduled times in the pre-interventional period and after finishing the intervention period.

The DPP is a flexible, individualized program that gives each participant some freedom to follow their preferences according to individual needs. For example, sedentary participants at the beginning of the intervention are advised to consistently increase their physical activity from their inactivity, with the eventual goal of doing 150 minutes per week of moderate aerobic exercise by the end of the intervention, rather than mandating a particular predefined amount of exercise in the first week.

The health-coach will monitor attendance of the weekly teaching sessions, offering make- up teaching for missed sessions on an individual basis while encouraging individual participation in their family's efforts at adhering to the program. The health coach will also monitor individual progress towards the goals of increasing physical activity and making healthier dietary choices. Each participant will have access to help, advice, and support from the health coach during the intervention period.

Participants with comorbid conditions will be instructed to continue any individual treatment plans under the ongoing supervision of their primary physician and any specialists; they will be advised that any medications they take may need to be adjusted by the preexisting care team in case the anticipated weight loss results in significant changes in blood sugar or blood pressure. The only criteria for stopping the intervention will be withdrawal of participant consent.

Prior studies done in the UAE have been hampered by low levels of retention of participants during the study period. Similar challenges exist for this study, as loss to follow up is quite common in the investigatory team's own experience. The therapeutic relationship between the health coach and family is the primary measure that will improve adherence and participant retention. To this end, the investigators have selected a health coach who speaks Arabic, has worked in the UAE for over thirty years as a medical interpreter within the government health system, is knowledgeable in local customs and practices, and has a degree in psychology. The health coach also has experience in working with this patient population as the outpatient clinical care coordinator, who arranges follow up appointments and is responsible for contacting patients with reminders.

Outcomes Primary outcome measure The primary outcome measure is the difference between the participant's pre- and post-intervention weight. This conforms with the American Diabetes Association guidelines on the management of diabetes which states that weight reduction of even 5% from baseline is associated with a clinically significant improvement in glycemic control and cardiovascular risk. Weight reduction is also a popular goal which is easily measured and analyzed.

Secondary outcome measures

Secondary measures include the absolute and relative change pre- and post-intervention in:

* Systolic blood pressure
* Diastolic blood pressure
* Hemoglobin A1c
* Total cholesterol
* HDL cholesterol
* LDL cholesterol
* Triglycerides

Participant timeline The primary and secondary measures will be assessed before intervention in eligible family members according to the randomized schedule. The sixteen sessions will then be delivered with coaching in between sessions. Afterthe final session, the participant will have repeat measurements of the primary and secondary measures.

Sample size Clusters will be analyzed for inter- and intracluster correlation. Assuming that the fluctuation in mean weight (i.e. the standard deviation) is 3.5%, we would need four clusters in each arm, for a total of eight clusters to achieve a power of 80% and a significance level of 5% for a two-armed parallel cluster randomized design. Since the selected stepped- wedge cluster design is more efficient than a parallel design, this sample size should be adequate to begin with.

Once four clusters have completed the intervention, an interim analysis will be performed and the required sample size will be re-calculated on the basis of observed fluctuations in parameters. If this leads to the conclusion that more than 300 patients are required to detect a statistical significance in the primary outcome, the study will be stopped as the relative benefit is judged to be clinically insignificant.

Recruitment Participants will be recruited from patients presenting to Kanad Hospital based on the eligibility criteria, as well as participant interest and consent. Screening and recruitment will continue until the required sample size is achieved or the grant expires, whichever occurs first.

Allocation Due to the limited resources available, it is not possible to perform a parallel cluster randomized trial. In addition, variation in the size of the family units makes such a family-to-family comparison impractical. Therefore, a stepped-wedge cluster randomized design was selected.

If a positive trial result is obtained, additional funding and health coaches could be requested to allow for further study.

Blinding Due to the nature of the intervention, it is impossible to blind the participants in the interventional and control arms, as the participants in the interventional period will receive teaching and coaching in family meetings, whereas individuals in the pre-intervention period will be having individual appointments with the dietician without health coaching support and without being supplied activity trackers for personal use.

Data collection Primary outcome Weight: Increased weight is associated risk factors for cardiovascular disease. The American Diabetes Association guidelines for the management of prediabetes and diabetes recommend lifestyle changes to achieve a weight reduction of 7% in obese and overweight patients. Weight will be measured in clinic at scheduled times before and after the intervention. The clinic which will provide biometric and lab measurements has appropriate protocols for the calibration of the scales used in the clinic according to the manufacturers' specifications. The staff nurse measures the patient's weight at each clinic visit, and this data is stored in the electronic medical record. Each cluster will be given a scale within the home for weight measurements, which will allow the health coach to monitor participants' progress in weight reduction. If progress is less than expected, individualized support will be offered. The relationship between the health-coach and study participants is anticipated to increase retention in the interventional period.

In cases of study discontinuation or withdrawal, the data for the intervention participants will be classified under intention to treat.

Secondary outcomes The secondary outcomes of blood pressure, hemoglobin A1c, and lipid parameters will also be obtained in the clinic at scheduled times prior to and after completing the intervention. The blood pressure is measured by an automated sphygmomanometer which undergoes routine calibration. A single accredited laboratory will perform the analyses of the blood samples.

Method of analysis A mixed random and fixed effects linear model will be utilized where the parameters measured at the end of each period will be the dependent outcome values. These will be analyzed so values will be fixed covariables, as well as whether the episode was an "post-intervention" or "pre-intervention" episode. Random effects are the family units.

Episodes after the post-intervention episode will be excluded from the main analysis and used to explore the persistence of intervention effects.

Data monitoring Data will be shared with the Kanad Hospital Research Ethics Committee (KHREC), which is independent of the investigators and the University of the United Arab Emirates. KHREC is responsible for ensuring the ethical nature of all research involving human subjects within Kanad Hospital and stopping any study that has significant concerns regarding ethics or participant safety. Interim analyses will be supplied confidentially to KHREC along with any additional requested data. Currently, an interim analysis is scheduled when 50% of the calculated sample size (4 family clusters) is enrolled.

Due to the benign nature of the intervention and the stringent oversight supplied by KHREC, a dedicated Data Monitoring Committee was not required for this study.

Harms Because this study involves lifestyle modification only, no significant risk of harm is anticipated. Each study participant will continue separately under the care of their primary care physician. As part of the informed consent, each participant is counselled that any medications are taken may need to be adjusted due to weight loss.

An adverse event, for the purposes of the study, will be defined as any event with a potentially or actually negative effect on the participant's health. The most likely adverse event would be hypoglycemia in those participants who may be taking certain medications for diabetes. The investigators decided to include patients on medications for diabetes in order to increase the generalizability of this study and to assess the real world effect of the package of interventions on patients who are overweight or obese. The potential for adverse effects is included in the informed consent form, along with the contact information for the principal investigator (JK).

The health coach is aware of the symptoms of hypoglycemia, and which medications potentially place participants at increased risk. The coach will educate any participants on these medications on how to initially manage hypoglycemia, as well as the need to follow up with the primary physician or emergency services after the initial management phase.

At each session, the participants who are present will be asked by the health coach if any problems were encountered, and any potential adverse events will be reported to the principal investigator for further evaluation. In significant cases, a report including the nature of the adverse event, severity, and potential causes will be sent to KHREC. Severe events or events that cannot be attributed to other causes other than the study intervention will be reported to the Ethics Committee within 24 hours.

Consent Eligible individuals will be asked to invite family members to enroll together in the study. These family members will then undergo screening for eligibility as well. Interested individuals who meet the eligibility criteria will then read the informed consent either in English or Arabic. Any questions or concerns will be addressed by one of the investigators in either English or Arabic, with translation as needed. All of the investigators are medical doctors and experienced researchers. Once this process is completed, and all questions and concerns are addressed, those who are interested in participating will be enrolled upon signing the informed consent form in the appropriate language (English or Arabic). One of the inclusion criteria is the ability of each potential participant to give informed consent for enrollment in the trial; if there is any concern on the investigators' part regarding the capacity of that individual to give consent, that person will be excluded from the study.

Confidentiality The biometric and lab data will be stored as usual in the participants' electronic medical record, which is access restricted, password protected, and otherwise safeguarded by the information technology team of Kanad Hospital. Participants' data will not be released outside of the study without individual written permission, except as requested for monitoring purposes by KHREC or as legally required by local or national government authorities.

Access to data Only those investigators who perform clinical duties at Kanad Hospital (AK, KC) will have access to the original pre and post-intervention biometric and lab data via the participants' electronic medical record. Once the data has been de-identified, all of the investigators will have access to de-identified data. The health coach and investigators will have access to the data supplied by each participant on a weekly basis, which includes but is not limited to weight, caloric intake, minutes and type of exercise, and correspondence. Access will be discontinued after the aggregate data has been analyzed and published.

Ancillary and post-trial care All Emiratis who are eligible for this study have comprehensive health insurance which will cover, at no cost to the participant, any needed medical care. No additional compensation is anticipated or required due to benign nature of the intervention.

Should this study provide evidence of a clinically significant benefit to those who underwent the study intervention, the age and gender matched controls will be contacted at the conclusion of the study and invited to receive the same intervention at the discretion of Kanad Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Emirati citizenship
* Age 18 years or older
* Able to give informed consent for study participation
* BMI 25 or greater

Exclusion Criteria:

* Current or planned use of weight-loss pharmacotherapy;
* Recent (within 6 months) bariatric surgery;
* Current diagnosis of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Weight | 16 weeks
  Weight (change from enrollment to end of intervention)

SECONDARY OUTCOMES:
Systolic blood pressure | 16 weeks
  Systolic blood pressure (change from enrollment to end of intervention)
Diastolic blood pressure | 16 weeks
  Diastolic blood pressure (change from enrollment to end of intervention)
Hemoglobin A1c | 16 weeks
  Hemoglobin A1c (change from enrollment to end of intervention)
Total cholesterol | 16 weeks
  Total cholesterol (change from enrollment to end of intervention)
HDL cholesterol | 16 weeks
  HDL cholesterol (change from enrollment to end of intervention)
LDL cholesterol | 16 weeks
  LDL cholesterol (change from enrollment to end of intervention)
Triglycerides | 16 weeks
  Triglycerides (change from enrollment to end of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey K King, MD, Principal Investigator — Assistant professor
Locations (1):
- Kanad Hospital, Al Ain City, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
For privacy reasons, identifiable health information cannot be shared.

REFERENCES:
- [Background] Loney T, Aw TC, Handysides DG, Ali R, Blair I, Grivna M, Shah SM, Sheek-Hussein M, El-Sadig M, Sharif AA, El-Obaid Y. An analysis of the health status of the United Arab Emirates: the 'Big 4' public health issues. Glob Health Action. 2013 Feb 5;6:20100. doi: 10.3402/gha.v6i0.20100. PMID 23394856
- [Background] Afshin A, Micha R, Khatibzadeh S, Fahimi S, Shi P, Powles J, Singh G, Yakoob MY, Abdollahi M, Al-Hooti S, Farzadfar F, Houshiar-Rad A, Hwalla N, Koksal E, Musaiger A, Pekcan G, Sibai AM, Zaghloul S, Danaei G, Ezzati M, Mozaffarian D; 2010 Global Burden of Diseases, Injuries, and Risk Factors Study: NUTRItrition and ChrOnic Diseases Expert Group (NUTRICODE), and Metabolic Risk Factors of ChrOnic Diseases Collaborating Group. The impact of dietary habits and metabolic risk factors on cardiovascular and diabetes mortality in countries of the Middle East and North Africa in 2010: a comparative risk assessment analysis. BMJ Open. 2015 May 20;5(5):e006385. doi: 10.1136/bmjopen-2014-006385. PMID 25995236
- [Background] Ratner R, Goldberg R, Haffner S, Marcovina S, Orchard T, Fowler S, Temprosa M; Diabetes Prevention Program Research Group. Impact of intensive lifestyle and metformin therapy on cardiovascular disease risk factors in the diabetes prevention program. Diabetes Care. 2005 Apr;28(4):888-94. doi: 10.2337/diacare.28.4.888. PMID 15793191
- [Background] Diabetes Prevention Program Outcomes Study Research Group; Orchard TJ, Temprosa M, Barrett-Connor E, Fowler SE, Goldberg RB, Mather KJ, Marcovina SM, Montez M, Ratner RE, Saudek CD, Sherif H, Watson KE. Long-term effects of the Diabetes Prevention Program interventions on cardiovascular risk factors: a report from the DPP Outcomes Study. Diabet Med. 2013 Jan;30(1):46-55. doi: 10.1111/j.1464-5491.2012.03750.x. PMID 22812594
- [Background] Diabetes Prevention Program Research Group. Long-term effects of lifestyle intervention or metformin on diabetes development and microvascular complications over 15-year follow-up: the Diabetes Prevention Program Outcomes Study. Lancet Diabetes Endocrinol. 2015 Nov;3(11):866-75. doi: 10.1016/S2213-8587(15)00291-0. Epub 2015 Sep 13. PMID 26377054
- [Background] Nathan DM, Bennett PH, Crandall JP, Edelstein SL, Goldberg RB, Kahn SE, Knowler WC, Mather KJ, Mudaliar S, Orchard TJ, Temprosa M, White NH; Research Group. Does diabetes prevention translate into reduced long-term vascular complications of diabetes? Diabetologia. 2019 Aug;62(8):1319-1328. doi: 10.1007/s00125-019-4928-8. Epub 2019 Jul 4. PMID 31270584
- [Background] Al-Kaabi J, Al-Maskari F, Saadi H, Afandi B, Parkar H, Nagelkerke N. Physical activity and reported barriers to activity among type 2 diabetic patients in the United arab emirates. Rev Diabet Stud. 2009 Winter;6(4):271-8. doi: 10.1900/RDS.2009.6.271. Epub 2009 Dec 30. PMID 20043039
- [Derived] King JK, Sheek-Hussein M, Nagelkerke NJD, Kieu A, Al-Shamsi S, Nauman J, Hoque N, Govender RD, ElBarazi I, Crawford K. Emirates Heart Health Project (EHHP): A protocol for a stepped-wedge family-cluster randomized-controlled trial of a health-coach guided diet and exercise intervention to reduce weight and cardiovascular risk in overweight and obese UAE nationals. PLoS One. 2023 Apr 10;18(4):e0282502. doi: 10.1371/journal.pone.0282502. eCollection 2023. PMID 37036843